CLINICAL TRIAL: NCT04429165
Title: RetroBRACE II: Clinical and Functional Outcomes 2 Years After ACL Repair and InternalBrace Ligament Augmentation in Comparison With ACL Reconstruction - Considering Socioeconomic Aspects and Return to Work
Brief Title: Clinical and Functional Outcomes 2 Years After ACL Repair and InternalBrace Ligament Augmentation in Comparison With ACL Reconstruction
Acronym: RetroBRACE II
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00551; ch20Rikli
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Injury of the Anterior Cruciate Ligament (ACL)
Keywords: ACL rupture; primary ACL repair; ACL reconstruction using autologous hamstring tendons; InternalBraceTM Ligament Augmentation
MeSH Terms: interventions — prolyl-proline; Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACL reconstruction: ACL reconstruction using an autologous hamstring tendon
  Interventions: Other: collection of Patient Reported Outcome (PRO) data; Other: collection of anthropometric and clinical functional data; Other: gait analysis
- control group: knee-healthy, age-matched subjects as a control group
  Interventions: Other: collection of Patient Reported Outcome (PRO) data; Other: collection of anthropometric and clinical functional data; Other: gait analysis

INTERVENTIONS:
Other: collection of Patient Reported Outcome (PRO) data — collection of Patient Reported Outcome (PRO) data by questionnaires
Other: collection of anthropometric and clinical functional data — collection of anthropometric and clinical functional data including range of motion (ROM), isokinetic muscle strength, joint position sense, single leg balance ability, and muscle activity
Other: gait analysis — gait analysis in a motion capture volume on a walkway including force plates and on a treadmill with pressure plates, while 3D kinematics and kinetics, pressure and electromyographic (EMG) data will be recorded

SUMMARY:
The aim of this study is to assess the clinical, biomechanical and functional outcome 2 years after anterior cruciate ligament (ACL) repair and InternalBraceTM augmentation now in direct comparison to ACL reconstruction and to identify potential deficits compared to the contralateral healthy side as well as with a knee-healthy age-matched collective. In addition, socio-economic aspects such as return to work and sports and treatment cost will be compared between both techniques.

DETAILED DESCRIPTION:
Injury of the anterior cruciate ligament (ACL) is one of the most common injuries of the knee. Since May 2016, patients with proximal ruptures of the ACL have been treated with direct repair and InternalBraceTM Ligament Augmentation at the University Hospital of Basel.

The remodelling of hamstring grafts used for ACL reconstruction is completed at the earliest 2 years after the surgery. The aim of this study is to assess the clinical, biomechanical and functional outcome 2 years after anterior cruciate ligament (ACL) repair and InternalBraceTM augmentation now in direct comparison to ACL reconstruction and to identify potential deficits compared to the contralateral healthy side as well as with a knee-healthy age-matched collective. In addition, socio-economic aspects such as return to work and sports and treatment cost will be compared between both techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients: 2 years since ACL reconstruction with autologous hamstring tendon
* Control subjects: no previous injury to the meniscus or the ligament apparatus of the knee

Exclusion Criteria:

* BMI > 35 kg / m2
* neuromuscular diseases that affect lower limb movement
* Inability to give informed consent
* Patients: previous injury or surgical treatment of the opposite side within the past 2 years and the injured leg within the past 6 months; other pathologies that affect the mobility of the knee

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who underwent ACL reconstruction using an autologous hamstring tendon between 03/18 and 04/20 at University Hospital Basel.
  30 age-matched control subjects without previous history of knee injury and/or surgery will be included for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Range of Motion (ROM) of the knee | at baseline (2 years after surgery)
  Range of Motion (ROM) of the knee
Isokinetic muscle strength | approx. 30 minutes at baseline (2 years after surgery)
  Isokinetic muscle strength will be measured bilaterally using a dynamometer (Biodex System 4 Pro: Biodex Medical Systems, Shirley, NY, USA). The maximum isokinetic flexion and extension torques will be measured on the knee between full extension and 90° flexion at a movement speed of 60°/s (5 repetitions) and 240°/s (15 repetitions). Maximum torques will be recorded for each direction of movement and normalized to body weight.
Proprioception (joint position sense) | approx. 30 minutes at baseline (2 years after surgery)
  Proprioception will be measured bilaterally with a dynamometer (Biodex System 4 Pro: Biodex Medical Systems, Shirley, NY, USA) using an active joint position sense protocol. The participants will be positioned on the dynamometer with knee and hip angles of 90°. They will then actively stretch their knees up to target angles of 60° or 30° flexion. Subjects will be asked to remember this position and then stretch their knees from a starting position of 90° flexion and, as soon as they think they have reached the target angle, push a stop button. The deviation between the perceived angle and the actual target angle will be calculated.
Gait analysis | approx. 60 minutes at baseline (2 years after surgery)
  Gait analysis performed on a treadmill with an integrated pressure plate and a walkway with two integrated force plates. Kinematic and EMG data collected using a 9-camera Vicon system and a 12-channel EMG system. To measure 3D joint angles, reflective markers will be attached to defined anatomical locations on the pelvis and legs.10 Bipolar surface electrodes will be attached bilaterally to the glutaeus medius, vastus medialis and lateralis, semitendinosus, tibialis anterior and gastrocnemius medialis muscles according to the SENIAM project (Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles). Study participants walk at self-selected speed. In addition, patients walk on treadmill at a self-selected speed, at a speed of 1.2 m/s and to run at self-selected speed and if possible at 2.2m/s. Kinematic and kinetic, EMG and pressure data recorded for all testing conditions.
Postural stability | at baseline (2 years after surgery)
  The stability of posture and balancing will be determined by the variability of movement in the horizontal plane and the length of the pressure line during two 30-second single- leg stands (on solid surface and on foam surface) on a force plate (Kistler 9260AA6, Kistler AG, Winterthur, Switzerland; sampling frequency, 2400 Hz) and mathematical calculations
Functional activity score to determine the ability "return to activity" | at baseline (2 years after surgery)
  Functional activity tests include the Y-balance test, single-leg jump for distance, side jumps for time (30 seconds) and precision over a distance of 40 cm (side hop). The quantity of movement of these functional scores will be calculated.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | at baseline (2 years after surgery)
  questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee Problems.
International Knee Documentation Committee (IKDC) | at baseline (2 years after surgery)
  The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function
Tegner Activity Score | at baseline (2 years after surgery)
  Tegner activity level scale is a graduated list of activities of daily living, recreation, and competitive sports. A score of 0 represents sick leave or disability pension because of knee problems, whereas a score of 10 corresponds to participation in national and international elite competitive sports.
EuroQoL-5D-5L (EQ 5D 5L) | at baseline (2 years after surgery)
  EQ-5D-5L questionnaire measuring generic health Status; descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 55555 (having extreme problems in all dimensions).
ACL- RSI Score | at baseline (2 years after surgery)
  The ALC-RSI measures the patient's understanding of his knee. It comprises 12 questions with a score of 1 to 10 for each. It is considered that for a normal population without knee condition, the score is between 80 and 90%
Time to return to work | at baseline (2 years after surgery)
  Socioeconomic aspect: time to return to work
Time to return to sports | at baseline (2 years after surgery)
  Time to return to sports

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mueller, Dr. med., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Buhl L, Muller S, Nuesch C, Boyer KA, Casto E, Mundermann A, Egloff C. Ambulatory knee biomechanics and muscle activity 2 years after ACL surgery: InternalBraceTM-augmented ACL repair versus ACL reconstruction versus healthy controls. BMC Musculoskelet Disord. 2023 Oct 4;24(1):785. doi: 10.1186/s12891-023-06916-7. PMID 37794432
- [Derived] Buhl L, Muller S, Nuesch C, Pagenstert G, Mundermann A, Egloff C. Functional leg performance 2 years after ACL surgery: a comparison between InternalBrace-augmented repair versus reconstruction versus healthy controls. J Orthop Traumatol. 2023 Sep 21;24(1):52. doi: 10.1186/s10195-023-00723-5. PMID 37735271
- [Derived] Muller S, Buhl L, Nuesch C, Pagenstert G, Mundermann A, Egloff C. Favorable Patient-Reported, Clinical, and Functional Outcomes 2 Years After ACL Repair and InternalBrace Augmentation Compared With ACL Reconstruction and Healthy Controls. Am J Sports Med. 2023 Oct;51(12):3131-3141. doi: 10.1177/03635465231194784. Epub 2023 Sep 7. PMID 37675973
- [Derived] Muller S, Buhl L, Nuesch C, Pagenstert G, Mundermann A, Egloff C. RetroBRACE: clinical, socioeconomic and functional-biomechanical outcomes 2 years after ACL repair and InternalBrace augmentation in comparison to ACL reconstruction and healthy controls-experimental protocol of a non-randomised single-centre comparative study. BMJ Open. 2022 Feb 1;12(2):e054709. doi: 10.1136/bmjopen-2021-054709. PMID 35105587